CLINICAL TRIAL: NCT00101595
Title: A Phase II Study of BMS-354825 in Subjects With Lymphoid Blast Phase Chronic Myeloid Leukemia or Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia Resistant to or Intolerant of Imatinib Mesylate
Brief Title: Dasatinib (BMS-354825) in Subjects With Lymphoid Blast Phase Chronic Myeloid Leukemia or Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA180-015; NCT00110097 (obsolete NCT alias)
Record Dates: First submitted 2005-01-12; First posted 2005-01-13 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Chronic Myeloid Leukemia; Leukemia, Lymphoblastic, Acute, Philadelphia-positive
Keywords: Lymphoid blast phase chronic myeloid leukemia; Philadelphia chromosome positive acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Tablets, Oral, 70 mg, twice daily, Until disease progression or untolerable toxicity, switch to the roll-over study or study closure
  Other Names: BMS-354825; Sprycel

SUMMARY:
The purpose of this clinical research study is to learn if BMS-354825 will have activity as defined by hematologic responses in subjects with lymphoid blast phase chronic myeloid leukemia (CML) and Philadelphia chromosome positive acute lymphoblastic leukemia with primary or acquired resistance to imatinib mesylate.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Philadelphia chromosome positive (Ph+) (BCR/ABL+) lymphoid blast phase chronic myeloid leukemia whose disease has primary or acquired hematologic resistance to imatinib mesylate or who are intolerant of imatinib mesylate.
* Subjects who are considered to have lymphoid blast phase CML if they meet at least one of the following criteria: *30% lymphoid blasts in peripheral blood or bone marrow. *Extramedullary infiltrates of leukemic cells (other than in spleen or liver) with peripheral blood lymphoid blast morphology.
* ECOG performance status score 0-2.
* Adequate hepatic function defined as: *Total bilirubin less than or equal to 2.0 times the institutional upper limit of normal; *alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 2.5 times the institutional upper limit of normal.
* Adequate renal function defined as: *serum creatinine less than or equal to 1.5 times the institutional upper normal limit.
* Men and women, 18 years of age or older.
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for a period of at least 1 month before and at least 3 months after the study in such a manner that the risk of pregnancy is minimized. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IC/L or equivalent units of HCG) within 72 hours prior to the start of study medication.

Exclusion Criteria:

* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period of at least 1 month before and for at least 3 months after completion of the study medication.
* WOCBP using a prohibited contraceptive method (not applicable).
* Women who are pregnant or breastfeeding.
* Women with a positive pregnancy test on enrollment or prior to study drug administration.
* Men whose sexual partners are WOCBP, who are unwilling or unable to use an acceptable method to avoid pregnancy of his partner for the entire study period and for at least 3 months after completion of study medication.
* Subjects who are eligible and willing to undergo transplantation during the screening period.
* A serious uncontrolled medical disorder or active infection that would impair the ability of the subject to receive protocol therapy.
* Demential or altered mental status that would prohibit the understanding or rendering of informed consent.
* History of significant bleeding disorder unrelated to CML.
* Concurrent incurable malignancy other than CML.
* Evidence of organ dysfunction or digestive dysfunction that would prevent administration of study therapy.
* Subjects who received any of the following:

  * imatinib mesylate within 7 days;
  * interferon or cytarabine within 14 days;
  * a targeted small molecule anti-cancer agent within 14 days;
  * any other investigational or antineoplastic agent other than hydroxyurea or anagrelide within 28 days before starting treatment with BMS-354825.
* Subjects currently taking drugs that are generally accepted to have a risk of causing Torsades de Pointes.
* Subjects taking medications that irreversibly inhibit platelet function.
* Prior therapy with BMS-354825.
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2005-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Major and overall hematologic response rates | throughout the study

SECONDARY OUTCOMES:
Durability of hematologic response and time to hematologic response (major and overall) | throughout the study
Assess cytogenetic and molecular responses | throughout the study
Measure minor hematologic response rate in the imatinib resistant group | throughout the study
Explore the role of BCR-ABL mRNA expression and point mutations in the BCR-ABL gene | throughout the study
Measure the heath-related QOL using FACT-G | throughout the study
To assess safety and tolerability of dasatinib | throughout the study
Population PK | first month

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (60):
- United States (18):
  - Local Institution, Birmingham, Alabama
  - Local Institution, Anaheim, California
  - Local Institution, Los Angeles, California
  - Local Institution, Stanford, California
  - Local Institution, Vallejo, California
  - Local Institution, Jacksonville, Florida
  - Local Institution, Tampa, Florida
  - Local Institution, Atlanta, Georgia
  - Local Institution, Chicago, Illinois
  - Local Institution, Kansas City, Kansas
  - Local Institution, Boston, Massachusetts
  - Local Institution, St Louis, Missouri
  - Local Institution, Hackensack, New Jersey
  - Local Institution, New York, New York
  - Local Institution, Portland, Oregon
  - Local Institution, Pittsburgh, Pennsylvania
  - Local Institution, Nashville, Tennessee
  - Local Institution, Houston, Texas
- Argentina (2):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
- Local Institution, St Leonards, New South Wales, Australia
- Local Institution, Vienna, Austria
- Belgium (3):
  - Local Institution, B-Leuven
  - Local Institution, Edegem
  - Local Institution, Yvoir
- Brazil (2):
  - Local Institution, São Paulo, São Paulo
  - Local Institution, Campinas
- Canada (2):
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
- Local Institution, Aarhus, Denmark
- Local Institution, Helsinki, Finland
- France (7):
  - Local Institution, Lille
  - Local Institution, Lyon
  - Local Institution, Nantes
  - Local Institution, Paris
  - Local Institution, Pessac
  - Local Institution, Poitiers
  - Local Institution, Strasbourg
- Germany (4):
  - Local Institution, Frankfurt am Main
  - Local Institution, Hamburg
  - Local Institution, Mainz
  - Local Institution, Mannheim
- Local Institution, Ramat Gan, Israel
- Italy (3):
  - Local Institution, Bologna
  - Local Institution, Orbassano
  - Local Institution, Roma
- Netherlands (2):
  - Local Institution, Nijmegen
  - Local Institution, Rotterdam
- Local Institution, Trondheim, Norway
- Local Institution, Lima, Lima Province, Peru
- South Korea (2):
  - Local Institution, Kyunggi-Do
  - Local Institution, Seoul
- Sweden (5):
  - Local Institution, Gothenburg
  - Local Institution, Lund
  - Local Institution, Stockholm
  - Local Institution, Umeå
  - Local Institution, Uppsala
- Local Institution, Basel, Switzerland
- United Kingdom (2):
  - Local Institution, Glasgow, Central
  - Local Institution, London, Greater London

REFERENCES:
- [Background] Cortes J, Rousselot P, Kim DW, Ritchie E, Hamerschlak N, Coutre S, Hochhaus A, Guilhot F, Saglio G, Apperley J, Ottmann O, Shah N, Erben P, Branford S, Agarwal P, Gollerkeri A, Baccarani M. Dasatinib induces complete hematologic and cytogenetic responses in patients with imatinib-resistant or -intolerant chronic myeloid leukemia in blast crisis. Blood. 2007 Apr 15;109(8):3207-13. doi: 10.1182/blood-2006-09-046888. Epub 2006 Dec 21. PMID 17185463
- [Background] Ottmann O, Dombret H, Martinelli G, Simonsson B, Guilhot F, Larson RA, Rege-Cambrin G, Radich J, Hochhaus A, Apanovitch AM, Gollerkeri A, Coutre S. Dasatinib induces rapid hematologic and cytogenetic responses in adult patients with Philadelphia chromosome positive acute lymphoblastic leukemia with resistance or intolerance to imatinib: interim results of a phase 2 study. Blood. 2007 Oct 1;110(7):2309-15. doi: 10.1182/blood-2007-02-073528. Epub 2007 May 11. PMID 17496201
- [Background] Porkka K, Koskenvesa P, Lundan T, Rimpilainen J, Mustjoki S, Smykla R, Wild R, Luo R, Arnan M, Brethon B, Eccersley L, Hjorth-Hansen H, Hoglund M, Klamova H, Knutsen H, Parikh S, Raffoux E, Gruber F, Brito-Babapulle F, Dombret H, Duarte RF, Elonen E, Paquette R, Zwaan CM, Lee FY. Dasatinib crosses the blood-brain barrier and is an efficient therapy for central nervous system Philadelphia chromosome-positive leukemia. Blood. 2008 Aug 15;112(4):1005-12. doi: 10.1182/blood-2008-02-140665. Epub 2008 May 13. PMID 18477770